CLINICAL TRIAL: NCT03269695
Title: A PHASE 2A, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED STUDY TO EVALUATE THE EFFICACY, SAFETY, TOLERABILITY AND PHARMACOKINETICS OF PF-06687234 AS ADD-ON THERAPY TO INFLIXIMAB IN ACTIVE ULCERATIVE COLITIS SUBJECTS WHO ARE NOT IN REMISSION (BUILD UC)
Brief Title: Efficacy, Safety and Tolerability of PF-06687234 as Add-on Therapy to Infliximab in Active UC Subjects Not in Remission.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The Sponsor changed R&D strategy and priority.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B7581002; 2017-002108-28 (EudraCT Number); BUILD UC (Other: Alias Study Number)
Record Dates: First submitted 2017-08-30; First posted 2017-09-01 (Actual); Results first posted 2021-12-28 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-11

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PF-06687234 (Experimental): PF-06687234 subcutaneous (SC) weekly (QW) x 12 doses
  Interventions: Drug: PF-06687234
- Placebo (Placebo Comparator): PF-06687234 matched Placebo SC QW x 12 doses
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-06687234 — SC QW
  Other Names: Investigational product
  Arms: PF-06687234
Drug: Placebo — SC QW
  Other Names: PF-06687234 matched placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if PF-06687234 is effective and safe as add-on therapy to infliximab in subjects with active ulcerative colitis who are not in remission.

DETAILED DESCRIPTION:
This is a Phase 2a, double-blind, placebo-controlled, parallel group study in subjects with active ulcerative colitis and a non-remission (partial) response to infliximab. All enrolled subjects must have been on infliximab for a minimum of 14 weeks with last dose 8 weeks prior to the date of randomization. Subjects will be randomly assigned to 1 of 2 treatment arms (PF-06687234 or placebo) administered subcutaneously every week for a total of 12 doses. Blood, stool and tissue samples will be collected at various time points throughout the study to evaluate efficacy, safety, tolerability, pharmacokinetics and immunogenicity. Duration of participation for subjects will be approximately 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female subjects 18 years to 75 years of age and weight > 40 kg at the time of informed consent.
* A diagnosis of active UC (histologic) for 4 months.
* Subjects with active UC as defined by (via screening endoscopy) a total Mayo Score of 4 or more but 9 or less and an endoscopic subscore of 2.or more.
* UC extending at least 15 cm proximal to the anal verge at the time of the screening endoscopy.
* Must be on a stable dose 5-10 mg/kg of Remicade, Inflectra, or Remsima for a minimum of 14 weeks with no anticipation of need for change in infliximab treatment regimen throughout the study
* Male subjects able to father children and female subjects of childbearing potential and at risk for pregnancy must agree to use two methods of contraception (at least one of which is considered as highly effective) throughout the study and until the Week 16 visit

Exclusion Criteria:

* Subjects with a diagnosis or documented history of total colectomy and/or pouchitis, indeterminate colitis, microscopic colitis, ischemic colitis, infectious colitis, radiation colitis, and diverticular disease associated with colitis, or clinical findings suggestive of Crohn's disease.
* Subjects need for surgery or with major elective surgery scheduled during the study.
* Subjects with extensive colitis for at least 8 years who have not had a colonoscopy with surveillance biopsies within 2 years prior to baseline.
* Subjects with history of or at screening endoscopy, biopsy documented colonic dysplasia or neoplasia.
* Subjects who require infliximab dosing interval other than every 6 weeks or every 8 weeks.
* Subjects displaying clinical signs of fulminant colitis or toxic megacolon, with primary sclerosing cholangitis, known colonic stricture, history of colonic, small bowel obstruction or resection, with history of or current colonic or small bowel stoma.
* Cyclic neutropenia, thrombocytopenia, lymphopenia, leukopenia or history of chronic anemia.
* Presence of active enteric infection.
* Known history of human immunodeficiency virus (HIV) based on documented history with positive serological test, or positive HIV serologic test.
* Presence of transplanted organ.
* Anticipated need for any live vaccine.
* Class III or Class IV heart failure.
* Acute coronary syndrome and any history of cerebrovascular disease.
* Subjects with current, or a history of QT prolongation.
* Subjects receiving the following therapies within the designated time period:

  * >9 mg/day of oral budesonide or >20 mg/day of prednisone or equivalent within 2 weeks prior to baseline.
  * IV, IM or topical (rectal) treatment of 5-ASA or corticosteroid enemas within 2 weeks prior to baseline.
  * Anti integrin inhibitors within 14 weeks prior to baseline.
  * Any use of natalizumab.
  * Interferon therapy within 8 weeks prior to baseline.
  * Prior treatment with lymphocyte depleting therapies and alkylating agents.
  * Received selective B lymphocyte depleting agents within 1 year prior to baseline.
  * Receiving leukocyte apheresis, granulocyte apheresis, or plasma exchange within 6 months of baseline.
  * JAK inhibitors within 3 months prior to baseline.
  * Any investigational procedures(s) or product(s)30 days prior to baseline.
* History of sensitivity to heparin or heparin induced thrombocytopenia
* Known history of hypersensitivity, intolerance, or allergic reaction to PF-06687234 or any constituent of the IP.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2021-01-07 (Actual); Study Completion 2021-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (34):
- United States (14):
  - Dothan Surgery Center, Dothan, Alabama
  - Gut PC, dba Digestive Health Specialists of the Southeast, Dothan, Alabama
  - Emory Investigational Drug Services, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Emory University School of Medicine, Atlanta, Georgia
  - The Emory Clinic, Atlanta, Georgia
  - Chevy Chase Endoscopy Center, Chevy Chase, Maryland
  - MGG Group Co., Inc., Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - East Valley Endoscopy, Grand Rapids, Michigan
  - Eastside Endoscopy Center, Macomb, Michigan
  - Eastside Endoscopy Center, Saint Clair Shores, Michigan
  - Gastroenterology Associates of Western Michigan, PLC d.b.a. West Michigan Clinical Research Center, Wyoming, Michigan
  - Allegiance Research Specialists, Wauwatosa, Wisconsin
- Australia (6):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Eastern Health-Box Hill Hospital, Box Hill, Victoria
  - St. Vincent's Hospital, Melbourne, Fitzroy, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - St John Of God Health Care Inc. Trading as St. John of God Subiaco Hospital, Subiaco, Western Australia
- CHC Montlegia, Liège, Belgium
- Universitaetsklinikum Schleswig-Holstein Campus Kiel, Kiel, Germany
- The Chaim Sheba Medical Center, Ramat Gan, Israel
- Italy (3):
  - ASST Rhodense - Ospedale di Circolo di Rho, Rho, Milano
  - Azienda Ospedaliera di Padova, Padua
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma
- Saudi Arabia (3):
  - King Abdulaziz University Hospital, Jeddah
  - King Abdullah International Medical Research Center, Riyadh
  - King Khalid University Hospital, Riyadh
- Serbia (2):
  - CHC "Dr Dragisa Misovic-Dedinje", Belgrade
  - Clinical Hospital Center Zvezdara - Clinic for Gastroenterology and Hepatology, Belgrade
- South Korea (2):
  - The Catholic University of Korea, St. Vincent's Hospital, Gyeonggi-do
  - Kangbuk Samsung Hospital, Seoul
- Mersin Universitesi Tip Fakultesi Hastanesi, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7581002

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 46 participants were screened , of whom 20 were randomized and treated (10 participants each in the Placebo + Infliximab and PF-06687234 20 mg + Infliximab treatment groups). Fifteen participants completed the treatment.
Pre-assignment Details: Participants with active histologic Ulcerative Colitis (as defined by a total Mayo Score >= 4 but <=9 and an endoscopic subscore >=2) for >=4 months, and on a stable dose 5 to 10 mg/kg of Remicade, or protocol specified infliximab biosimilars for a minimum of 14 weeks prior to study entry with no anticipation of need for change in infliximab treatment regimen throughout the study were enrolled.
Groups:
- Placebo + Infliximab: Placebo for PF-06687234 was administered as subcutaneous injection on Day 1, Week 1 (Day 8), Week 2 (Day 15), Week 3 (Day 22), Week 4 (Day 29), Week 5 (Day 36), Week 6 (Day 43), Week 7 (Day 50), Week 8 (Day 57), Week 9 (Day 64), Week 10 (Day 71) and Week 11 (Day 78) for a total 12 doses. Remicade or protocol specified infliximab biosimilar was administered as an IV infusion on Day 1, Week 8 and Week 16 for a total of 3 doses for participants on infliximab every 8 weeks, and Day 1, Week 6, Week 12 and Week 18 for participants on infliximab every 6 weeks.
- PF-06687234 20 mg + Infliximab: PF-06687234 was administered as a 20 mg subcutaneous injection on Day 1, Week 1 (Day 8), Week 2 (Day 15), Week 3 (Day 22), Week 4 (Day 29), Week 5 (Day 36), Week 6 (Day 43), Week 7 (Day 50), Week 8 (Day 57), Week 9 (Day 64), Week 10 (Day 71) and Week 11 (Day 78) for a total 12 doses. Remicade or protocol specified infliximab biosimilar was administered as an IV infusion on Day 1, Week 8 and Week 16 for a total of 3 doses for participants on infliximab every 8 weeks, and Day 1, Week 6, Week 12 and Week 18 for participants on infliximab every 6 weeks.
Period: Overall Study
Arm/Group | Placebo + Infliximab | PF-06687234 20 mg + Infliximab
Started | 10 | 10
Treated | 10 | 10
Completed | 8 | 7
Not Completed | 2 | 3
Not completed — Adverse Event | 2 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of randomized treatment were included in the baseline analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Infliximab | PF-06687234 20 mg + Infliximab | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.6 (21.11) | 44.5 (12.44) | 44.6 (16.86)
Age, Continuous [Median (Full Range); unit: Years] | 44.5 [20 to 73] | 43.5 [20 to 64] | 43.5 [20 to 73]
Age, Customized [Count of Participants; unit: Participants]
  18-44 Years | 5 | 6 | 11
  45-64 Years | 2 | 4 | 6
  ≥ 65 Years | 3 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 7 | 6 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 8 | 8 | 16
  Asian | 2 | 2 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Modified Clinical Remission at Week 12 (Traditional Endoscopic Subscore <=1, Observed Cases)
Description: The Mayo score consists of 4 subscores (Endoscopic, stool frequency, rectal bleeding and Physician's global assessment [PGA]), each graded 0 to 3 with the higher score indicating more severe disease activity. Modified clinical remission is defined as a modified total Mayo Score (total Mayo score excluding the PGA subscore) <=2, no individual subscore >1, traditional endoscopic subscore <=1 (where mild friability was scored as of 1; moderate or severe friability was scored as 2) and rectal bleeding subscore=0. Participants with missing values were handled by observed case approach (the missing data were used as is). The percentage of participants achieving modified clinical remission was calculated based on the number of participants with observed data.
Time Frame: Week 12
Population: All participants who had received at least one dose of the randomized treatment (10 each for the Placebo + Infliximab arm and the PF-06687234 20mg + Infliximab arm).
Measure: Number (95% Confidence Interval); unit: Percentage of participants (%)
Arm/Group | Placebo + Infliximab | PF-06687234 20 mg + Infliximab
Number analyzed (Participants) | 10 | 10
Percentage of participants (%)
  Participants with missing data: number analyzed (Participants) | 2 | 3
  Participants with missing data | NA [NA to NA] — These participants did not have observed endoscopic data for the composite primary endpoint. | NA [NA to NA] — These participants did not have observed endoscopic data for the composite primary endpoint.
  Participants with observed data: number analyzed (Participants) | 8 | 7
  Participants with observed data | 12.5 [0.6 to 50.0] | 14.3 [0.7 to 55.0]
Statistical Analysis 1: Comparison: Placebo + Infliximab vs PF-06687234 20 mg + Infliximab; Test type: Superiority; p = 1.0000, Chan and Zhang (1999); Treatment difference = 1.8, 95% CI 2-sided [-41.0 to 47.2]

2. Primary Outcome: Percentage of Participants in Modified Clinical Remission at Week 12 (Traditional Mayo Endoscopic Subscore <=1, Treatment Failure Approach)
Description: The Mayo score consists of 4 subscores (Endoscopic, stool frequency, rectal bleeding and Physician's global assessment [PGA]), each graded 0 to 3 with the higher score indicating more severe disease activity. Modified clinical remission is defined as a modified total Mayo Score (total Mayo score excluding the PGA subscore) <=2, no individual subscore >1, traditional endoscopic subscore <=1 (where mild friability was scored as of 1; moderate or severe friability was scored as 2) and rectal bleeding subscore=0. Participants with missing values were handled by treatment failure approach (participants who had missing value for any reasons were considered as treatment failures).
Time Frame: Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants (%)
Arm/Group | Placebo + Infliximab | PF-06687234 20 mg + Infliximab
Number analyzed (Participants) | 10 | 10
Percentage of participants (%) | 10 [0.5 to 44.4] | 10 [0.5 to 44.4]
Statistical Analysis 1: Comparison: Placebo + Infliximab vs PF-06687234 20 mg + Infliximab; Test type: Superiority; p = 1.0000, Chan and Zhang (1999); Treatment difference = 0.0, 95% CI 2-sided [-37.0 to 37.0]

3. Primary Outcome: Percentage of Participants in Modified Clinical Remission at Week 12 (Modified Mayo Endoscopy Subscore = 0 or 1, Observed Cases)
Description: The Mayo score consists of 4 subscores (Endoscopic, stool frequency, rectal bleeding and Physician's global assessment), each graded 0 to 3 with the higher score indicating more severe disease activity. Modified clinical remission is defined as a modified total Mayo Score (total Mayo score excluding the PGA subscore) with endoscopic subscore = 0 or 1 (where any friability was scored as a mayo endoscopic subscore of 2), stool frequency subscore = 0 or 1, and rectal bleeding subscore = 0. Participants with missing values were handled by observed case approach (the missing data were used as is). The percentage of participants achieving modified clinical remission was calculated based on the number of participants with observed data.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants (%)
Arm/Group | Placebo + Infliximab | PF-06687234 20 mg + Infliximab
Number analyzed (Participants) | 10 | 10
Percentage of participants (%)
  Participants with missing data: number analyzed (Participants) | 2 | 3
  Participants with missing data | NA [NA to NA] — These participants did not have observed endoscopic data for the composite primary endpoint. | NA [NA to NA] — These participants did not have observed endoscopic data for the composite primary endpoint.
  Participants with observed data: number analyzed (Participants) | 8 | 7
  Participants with observed data | 0 [0.0 to 34.9] | 14.3 [0.7 to 55.4]
Statistical Analysis 1: Comparison: Placebo + Infliximab vs PF-06687234 20 mg + Infliximab; Test type: Superiority; p = 0.4700, Chan and Zhang (1999); Treatment difference = 14.3, 95% CI 2-sided [-23.8 to 57.9]

4. Primary Outcome: Percentage of Participants in Modified Clinical Remission at Week 12 (Modified Mayo Endoscopy Subscore = 0 or 1, Treatment Failure Approach)
Description: The Mayo score consists of 4 subscores (Endoscopic, stool frequency, rectal bleeding and Physician's global assessment [PGA]), each graded 0 to 3 with the higher score indicating more severe disease activity. Modified clinical remission is defined as a modified total Mayo Score (total Mayo score excluding the PGA subscore) with endoscopic subscore = 0 or 1 (where any friability was scored as a mayo endoscopic subscore of 2), stool frequency subscore = 0 or 1, and rectal bleeding subscore = 0. Participants with missing values were handled by treatment failure approach (participants who had missing value for any reasons were considered as treatment failures).
Time Frame: Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants (%)
Arm/Group | Placebo + Infliximab | PF-06687234 20 mg + Infliximab
Number analyzed (Participants) | 10 | 10
Percentage of participants (%) | 0 [0.0 to 26.7] | 10 [0.5 to 44.4]
Statistical Analysis 1: Comparison: Placebo + Infliximab vs PF-06687234 20 mg + Infliximab; Test type: Superiority; p = 0.5221, Chan and Zhang (1999); Treatment difference = 10.0, 95% CI 2-sided [-20.7 to 45.6]

5. Secondary Outcome: Percentage of Participants With Endoscopic Improvement at Week 12 ( Observed Cases)
Description: Endoscopic improvement is defined as a decrease of >=1 point in a modified endoscopic subscore (any friability is scored as 2) or an absolute endoscopy score of <=1 without friability. Participants with missing values were handled by observed case approach (the missing data were used as is). The percentage of participants achieving endoscopic improvement was calculated based on the number of participants with observed data.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants (%)
Arm/Group | Placebo + Infliximab | PF-06687234 20 mg + Infliximab
Number analyzed (Participants) | 10 | 10
Percentage of participants (%)
  Participants with missing data: number analyzed (Participants) | 2 | 3
  Participants with missing data | NA [NA to NA] — These participants did not have observed endoscopic data for this secondary endpoint. | NA [NA to NA] — These participants did not have observed endoscopic data for this secondary endpoint.
  Participants with observed data: number analyzed (Participants) | 8 | 7
  Participants with observed data | 25.0 [4.6 to 65.1] | 57.1 [22.5 to 87.1]
Statistical Analysis 1: Comparison: Placebo + Infliximab vs PF-06687234 20 mg + Infliximab; Test type: Superiority; p = 0.3166, Chan and Zhang (1999); Treatment difference = 32.1, 95% CI 2-sided [-23.7 to 74.1]

6. Secondary Outcome: Percentage of Participants With Endoscopic Improvement at Week 12 ( Treatment Failure Approach)
Description: Endoscopic improvement is defined as a decrease of >=1 point in a modified endoscopic subscore (any friability is scored as 2) or an absolute endoscopy score of <=1 without friability. Participants with missing values were handled by treatment failure approach (participants who had missing value for any reasons were considered as treatment failures).
Time Frame: Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants (%)
Arm/Group | Placebo + Infliximab | PF-06687234 20 mg + Infliximab
Number analyzed (Participants) | 10 | 10
Percentage of participants (%) | 20.0 [3.7 to 55.6] | 40.0 [15.0 to 73.3]
Statistical Analysis 1: Comparison: Placebo + Infliximab vs PF-06687234 20 mg + Infliximab; Test type: Superiority; p = 0.5234, Chan and Zhang (1999); Treatment difference = 20.0, 95% CI 2-sided [-22.9 to 58.5]

7. Secondary Outcome: Percentage of Participants Achieving Geboes Index Remission at Week 12 (Observed Cases)
Description: Geboes index is a structured six-grade classification system ordered as follows: 0, structural changes (sub-grade: 0-0.3); 1, chronic inflammatory infiltrate (sub-grade: 1-1.3); 2, lamina propria neutrophils and eosinophils (sub-grade: 2A-2B.3); 3, neutrophils in epithelium (sub-grade: 3-3.3); 4, crypt destruction (sub-grade: 4-4.3); and 5, erosion and ulceration (sub-grade: 5-5.4). The final index ranges from 0 to 5.4, with low score associated with no inflammation or less inflammation and high score associated with severe inflammation or ulceration. Geboes index remission was defined as Geboes index < 3 and Grade 3 < 3.1 at week 12. Participants with missing values were handled by observed case approach (the missing data were used as is). The percentage of participants achieving Geboes index remission was calculated based on the number of participants with observed data.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants (%)
Arm/Group | Placebo + Infliximab | PF-06687234 20 mg + Infliximab
Number analyzed (Participants) | 10 | 10
Percentage of participants (%)
  Participants with missing data: number analyzed (Participants) | 2 | 2
  Participants with missing data | NA [NA to NA] — These participants did not have observed endoscopic data for this secondary endpoint. | NA [NA to NA] — These participants did not have observed endoscopic data for this secondary endpoint.
  Participant with observed data: number analyzed (Participants) | 8 | 8
  Participant with observed data | 62.5 [28.9 to 88.9] | 37.5 [11.1 to 71.1]
Statistical Analysis 1: Comparison: Placebo + Infliximab vs PF-06687234 20 mg + Infliximab; Test type: Superiority; p = 0.7393, Chan and Zhang (1999); Treatment difference = -25.0, 95% CI 2-sided [-69.6 to 29.1]

8. Secondary Outcome: Change From Baseline in Robart's Histology Index at Week 12 (Observed Cases)
Description: Robart's histology index is based on the Geboes scores, and the final score is obtained by the summation of four main items (chronic inflammatory infiltrate level, lamina propria neutrophils, neutrophils in the epithelium, and erosion or ulceration), which are classified from 0 (no inflammation) to 3 (severe inflammation or ulceration), yielding a final score that ranges between 0 (no inflammation) and 33 (severe inflammation or ulceration). Participants with missing values were handled by observed case approach (the missing data were used as is).
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Placebo + Infliximab | PF-06687234 20 mg + Infliximab
Number analyzed (Participants) | 10 | 10
Scores on a scale
  Participants with missing data: number analyzed (Participants) | 2 | 2
  Participants with missing data | NA [NA to NA] — These participants did not have observed endoscopic data for this secondary endpoint. | NA [NA to NA] — These participants did not have observed endoscopic data for this secondary endpoint.
  Participants with observed data: number analyzed (Participants) | 8 | 8
  Participants with observed data | -12.96 [-20.60 to -5.32] | -7.16 [-14.81 to 0.48]
Statistical Analysis 1: Comparison: Placebo + Infliximab vs PF-06687234 20 mg + Infliximab; Test type: Superiority; p = 0.2705, ANCOVA; Least squares mean difference = 5.80, 95% CI 2-sided [-5.08 to 16.67]

9. Secondary Outcome: Percentage of Participants With a Clinical Response at Week 12 (Observed Cases)
Description: The Mayo score consists of 4 subscores (Endoscopic, stool frequency, rectal bleeding and Physician's global assessment [PGA]), each graded 0 to 3 with the higher score indicating more severe disease activity. Clinical response is defined with a decrease from baseline of at least 3 points in total Mayo score with at least 30% change, accompanied by at least one-point decrease or absolute score of 0 or 1 in rectal bleeding subscore. Participants with missing values were handled by observed case approach (the missing data were used as is).
Time Frame: Week 12
Population: All participants who have received at least one dose of the randomized treatment. The number of participants with observed data were 8 for the Placebo + Infliximab arm and 7 for PF-06687234 20mg + Infliximab arm. The percentage of participants achieving clinical response was calculated based on the number of participants with observed data.
Measure: Number (95% Confidence Interval); unit: Percentage of participants (%)
Arm/Group | Placebo + Infliximab | PF-06687234 20 mg + Infliximab
Number analyzed (Participants) | 10 | 10
Percentage of participants (%)
  Participants with missing data: number analyzed (Participants) | 2 | 3
  Participants with missing data | NA [NA to NA] — These participants did not have observed endoscopic data for this secondary endpoint. | NA [NA to NA] — These participants did not have observed endoscopic data for this secondary endpoint.
  Participants with observed data: number analyzed (Participants) | 8 | 7
  Participants with observed data | 37.5 [11.1 to 71.1] | 85.7 [44.6 to 99.3]
Statistical Analysis 1: Comparison: Placebo + Infliximab vs PF-06687234 20 mg + Infliximab; Test type: Superiority; p = 0.0732, Chan and Zhang (1999); Treatment difference = 48.2, 95% CI 2-sided [-4.4 to 84.7]

10. Secondary Outcome: Percentage of Participants With a Clinical Response at Week 12 (Treatment Failure Approach)
Description: The Mayo score consists of 4 subscores (Endoscopic, stool frequency, rectal bleeding and Physician's global assessment [PGA]), each graded 0 to 3 with the higher score indicating more severe disease activity. Clinical response is defined with a decrease from baseline of at least 3 points in total Mayo score with at least 30% change, accompanied by at least one-point decrease or absolute score of 0 or 1 in rectal bleeding subscore. Participants with missing values were handled by treatment failure approach (participants who had missing value for any reasons were considered as treatment failures).
Time Frame: Week 12
Population: All participants who have received at least one dose of the randomized treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants (%)
Arm/Group | Placebo + Infliximab | PF-06687234 20 mg + Infliximab
Number analyzed (Participants) | 10 | 10
Percentage of participants (%) | 30.0 [8.7 to 61.9] | 60.0 [26.7 to 85.0]
Statistical Analysis 1: Comparison: Placebo + Infliximab vs PF-06687234 20 mg + Infliximab; Test type: Superiority; p = 0.2633, Chan and Zhang (1999); Treatment difference = 30.0, 95% CI 2-sided [-18.4 to 69.2]

11. Secondary Outcome: Percentage of Participants With Change From Baseline in Derived Partial Mayo Score of <=2 With no Individual Subscore >1 at Weeks 2, 4, 8 and 12 (Observed Cases)
Description: The Mayo score is determined by the summation of 4 subscores (Endoscopic, stool frequency, rectal bleeding and Physician's global assessment [PGA]), each graded 0 (normal) to 3 (worst). Derived partial mayo score is defined as total Mayo score excluding the endoscopic subscore (stool frequency, rectal bleeding and PGA only), ranging from 0 (normal) to 9 (the most severe). The percentages of participants with change from baseline in derived partial Mayo score of <=2 with no individual subscore >1 at Weeks 2, 4, 8 and 12 were calculated for this endpoint. Participants with missing values were handled by observed case approach (the missing data were used as is). Generalized Linear Mixed Model (GLMM) was used with fixed effects of treatment, visit and treatment by visit interaction.
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: All participants who have received at least one dose of the randomized treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants (%)
Arm/Group | Placebo + Infliximab | PF-06687234 20 mg + Infliximab
Number analyzed (Participants) | 10 | 10
Percentage of participants (%)
  Week 2 | 50.0 [21.0 to 79.0] | 50.0 [21.0 to 79.0]
  Week 4 | 50.0 [21.0 to 79.0] | 60.0 [27.9 to 85.3]
  Week 8: number analyzed (Participants) | 9 | 9
  Week 8 | 62.5 [28.9 to 87.2] | 50.8 [20.9 to 80.1]
  Week 12: number analyzed (Participants) | 8 | 7
  Week 12 | 64.9 [29.8 to 89.0] | 64.8 [28.6 to 89.4]
Statistical Analysis 1: Comparison: Placebo + Infliximab vs PF-06687234 20 mg + Infliximab; At Week 2; Test type: Superiority; p = 1.0000, Generalized Linear Mixed Model; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.15 to 6.54]
Statistical Analysis 2: Comparison: Placebo + Infliximab vs PF-06687234 20 mg + Infliximab; At Week 4; Test type: Superiority; p = 0.6691, Generalized Linear Mixed Model; Odds Ratio (OR) = 1.50, 95% CI 2-sided [0.23 to 10.00]
Statistical Analysis 3: Comparison: Placebo + Infliximab vs PF-06687234 20 mg + Infliximab; At Week 8; Test type: Superiority; p = 0.6248, Generalized Linear Mixed Model; Odds Ratio (OR) = 0.62, 95% CI 2-sided [0.09 to 4.40]
Statistical Analysis 4: Comparison: Placebo + Infliximab vs PF-06687234 20 mg + Infliximab; At Week 12; Test type: Superiority; p = 0.9965, Generalized Linear Mixed Model; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.12 to 8.30]

12. Secondary Outcome: Serum Concentrations of PF-06687234 20 mg
Description: Samples for serum PF-06687234 concentration were collected approximately 30 minutes prior to dosing. Concentration values below the lower limit of quantification were excluded when calculating the geometric mean (geometric coefficient of variation).
Time Frame: Prior to dosing on Day 1 and at Weeks 1, 3, 7, 11, 12 (168 hours post dose) and 16
Population: All participants who received at least one dose of PF-06687234, had data on at least one PK concentration (above or equal to lower limit of quantification) and did not participate in PK substudy.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-06687234 20 mg + Infliximab
Number analyzed (Participants) | 10
ng/mL
  Day 1: number analyzed (Participants) | 0
  Week 1: number analyzed (Participants) | 0
  Week 3: number analyzed (Participants) | 2
  Week 3 | 0.4537 (42)
  Week 7: number analyzed (Participants) | 6
  Week 7 | 0.4494 (27)
  Week 11: number analyzed (Participants) | 3
  Week 11 | 0.4713 (2)
  Week 12: number analyzed (Participants) | 3
  Week 12 | 0.5140 (40)
  Week 16: number analyzed (Participants) | 0

13. Secondary Outcome: Percentage of Participants With the Development of Human Anti-Fusion Antibodies (HAFAs) and Neutralizing Antibodies (NAbs) Against PF-06687234
Description: Plasma samples were analyzed for anti PF-06687234, anti PF-06687234 IL-10 neutralizing antibody (AB) and anti PF-06687234 single chain variable fragment (scFv) neutralizing AB. Samples inadvertently analyzed were excluded.
Time Frame: At screening, Day 1, Weeks 3, 7, 11, 12 and 16 (prior to dosing)
Population: HAFA and NAb analyses were performed to characterize immunogenicity against PF-06687234, hence only participants who received at least one dose of PF-06687234 and with at least one post treatment HAFA determination were included.
Measure: Number; unit: Percentage of participants (%)
Arm/Group | PF-06687234 20 mg + Infliximab
Number analyzed (Participants) | 10
Percentage of participants (%)
  Anti PF-06687234 (Screening) | 0
  Anti PF-06687234 (Day 1) | 10.0
  Anti PF-06687234 (Week 3) | 30.0
  Anti PF-06687234 (Week 7): number analyzed (Participants) | 8
  Anti PF-06687234 (Week 7) | 50.0
  Anti PF-06687234 (Week 11): number analyzed (Participants) | 7
  Anti PF-06687234 (Week 11) | 28.6
  Anti PF-06687234 (Week 12): number analyzed (Participants) | 7
  Anti PF-06687234 (Week 12) | 28.6
  Anti PF-06687234 (Week 16): number analyzed (Participants) | 8
  Anti PF-06687234 (Week 16) | 12.5
  Anti PF-06687234 IL-10 neutralizing AB (Screening): number analyzed (Participants) | 0
  Anti PF-06687234 IL-10 neutralizing AB (Day 1): number analyzed (Participants) | 1
  Anti PF-06687234 IL-10 neutralizing AB (Day 1) | 0
  Anti PF-06687234 IL-10 neutralizing AB (Week 3): number analyzed (Participants) | 3
  Anti PF-06687234 IL-10 neutralizing AB (Week 3) | 0
  Anti PF-06687234 IL-10 neutralizing AB (Week 7): number analyzed (Participants) | 4
  Anti PF-06687234 IL-10 neutralizing AB (Week 7) | 0
  Anti PF-06687234 IL-10 neutralizing AB (Week 11): number analyzed (Participants) | 2
  Anti PF-06687234 IL-10 neutralizing AB (Week 11) | 0
  Anti PF-06687234 IL-10 neutralizing AB (Week 12): number analyzed (Participants) | 2
  Anti PF-06687234 IL-10 neutralizing AB (Week 12) | 0
  Anti PF-06687234 IL-10 neutralizing AB (Week 16): number analyzed (Participants) | 1
  Anti PF-06687234 IL-10 neutralizing AB (Week 16) | 0
  Anti PF-06687234 scFv neutralizing AB (Screening): number analyzed (Participants) | 0
  Anti PF-06687234 scFv neutralizing AB (Dany 1): number analyzed (Participants) | 1
  Anti PF-06687234 scFv neutralizing AB (Dany 1) | 0
  Anti PF-06687234 scFv neutralizing AB (Week 3): number analyzed (Participants) | 3
  Anti PF-06687234 scFv neutralizing AB (Week 3) | 0
  Anti PF-06687234 scFv neutralizing AB (Week 7): number analyzed (Participants) | 4
  Anti PF-06687234 scFv neutralizing AB (Week 7) | 50.0
  Anti PF-06687234 scFv neutralizing AB (Week 11): number analyzed (Participants) | 2
  Anti PF-06687234 scFv neutralizing AB (Week 11) | 0
  Anti PF-06687234 scFv neutralizing AB (Week 12): number analyzed (Participants) | 2
  Anti PF-06687234 scFv neutralizing AB (Week 12) | 0
  Anti PF-06687234 scFv neutralizing AB (Week 16): number analyzed (Participants) | 1
  Anti PF-06687234 scFv neutralizing AB (Week 16) | 0

14. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs; All Causalities)
Description: Treatment-emergent AEs are those with initial onset or that worsen in severity after the first dose of the study medication. All AEs in the table below were treatment-emergent AEs. An serious adverse event (SAE) is any untoward medical occurrence at any dose that: results in death; is life threatening (immediate risk of death); requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); results in congenital anomaly/birth defect; or that is considered to be an important medical event that may jeopardize the participant or may require intervention to prevent one of the other AE outcomes. Severe AEs were defined as AEs that interfered significantly with participant's usual function. Both SAEs and severe AEs were according to the investigator's assessment.
Time Frame: Baseline (Day 1) through and including a minimum of 28 calendar days after the last administration of the investigational products (22 weeks in total)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Infliximab | PF-06687234 20 mg + Infliximab
Number analyzed (Participants) | 10 | 10
Participants
  Participants with AEs | 8 | 9
  Participants with SAEs | 1 | 0
  Participants with severe AEs | 2 | 0
  Participants discontinued from study due to AEs | 0 | 0
  Participants discontinued study drug due to AEs and continued study | 2 | 1
  Participants with temporary discontinuation due to AEs | 1 | 1

15. Primary Outcome: Number of Participants With Treatment-Emergent AEs (Treatment Related)
Description: Treatment-emergent AEs are those with initial onset or that worsen in severity after the first dose of the study medication. All AEs in the table below were treatment-emergent AEs. An SAE is any untoward medical occurrence at any dose that: results in death; is life threatening (immediate risk of death); requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); results in congenital anomaly/birth defect; or that is considered to be an important medical event that may jeopardize the participant or may require intervention to prevent one of the other AE outcomes. Severe AEs were defined as AEs that interfered significantly with participant's usual function. Both SAEs and severe AEs were according to the investigator's assessment. Treatment-related AEs were also determined by the investigator.
Time Frame: as for outcome 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Infliximab | PF-06687234 20 mg + Infliximab
Number analyzed (Participants) | 10 | 10
Participants
  Participants with AEs | 1 | 7
  Participants with SAEs | 0 | 0
  Participants with severe AEs | 0 | 0
  Participants discontinued from study due to AEs | 0 | 0
  Participants discontinued study drug due to AEs and continued study | 1 | 0
  Participants with temporary discontinuation due to AEs | 0 | 0

16. Primary Outcome: Number of Participants With Laboratory Test Abnormalities Without Regard to Baseline Abnormality
Description: The laboratory tests as defined in the protocol, including hematology, chemistry, urinalysis and other, were performed. Baseline was defined as the last measurement prior to first dosing (Day 1).
Time Frame: From baseline through Week 16
Population: All participants with at least one observation of the given laboratory test while on study treatment or during lag time (10 each for the Placebo + Infliximab arm and the PF-06687234 20mg + Infliximab arm).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Infliximab | PF-06687234 20 mg + Infliximab
Number analyzed (Participants) | 10 | 10
Participants
  Hemoglobin (g/dL) < 0.8 x lower limit of normal (LLN) | 0 | 2
  Hematocrit (%) < 0.8 x LLN | 0 | 2
  Erythrocytes (10^6/mm^3) < 0.8 x LLN | 0 | 2
  Reticulocytes (10^3/mm^3) > 1.5 x upper limit of normal (ULN) | 0 | 1
  Reticulocytes/Erythrocytes (%) > 1.5 x ULN | 0 | 1
  Leukocytes (10^3/mm^3) > 1.5 x ULN | 0 | 1
  Lymphocytes (10^3/mm^3) < 0.8 x LLN | 2 | 2
  Lymphocytes/Leukocytes (%) < 0.8 x LLN | 1 | 4
  Neutrophils (10^3/mm^3) < 0.8 x LLN | 1 | 0
  Neutrophils (10^3/mm^3) > 1.2 x ULN | 0 | 2
  Neutrophils/Leukocytes (%) < 0.8 x LLN | 0 | 1
  Neutrophils/Leukocytes (%) > 1.2 x ULN | 0 | 2
  Basophils/Leukocytes (%) > 1.2 x ULN | 1 | 0
  Eosinophils (10^3/mm^3) > 1.2 x ULN | 0 | 1
  Eosinophils/Leukocytes (%) > 1.2 x ULN | 1 | 0
  Monocytes/Leukocytes (%) > 1.2 x ULN | 2 | 2
  Protein (g/dL) < 0.8 x LLN | 0 | 1
  Albumin (g/dL) < 0.8 x LLN | 1 | 1
  Creatinine (mg/dL) > 1.3 x ULN | 0 | 1
  Glucose (mg/dL) > 1.5 x ULN | 0 | 1
  Ketones (Scalar) >= 1 | 1 | 1
  Urine Protein (mg/dL) >= 1 | 1 | 1
  Urine Hemoglobin (Scalar) >= 1 | 3 | 3
  Leukocyte Esterase (Scalar) >= 1 | 4 | 3
  Hyaline Casts (/low-power field [LPF]) > 1: number analyzed (Participants) | 2 | 2
  Hyaline Casts (/low-power field [LPF]) > 1 | 0 | 2

17. Primary Outcome: Number of Participants With Categorical Vital Signs
Description: Single sitting blood pressure (BP), pulse rate, and temperature were measured. At Day 1 and Week 1, BP and pulse were collected approximately 30 minutes prior to dosing, approximately 30 minutes post dosing and approximately 1 hour post dosing. For participants with no safety issues (eg, severe injection site reactions, severe elevations BP and/or pulse), BP and pulse were collected approximately 30 minutes prior to dosing and approximately 30 minutes post dosing from Weeks 2-16. Vital signs were analyzed as per pre-specified categories.
Time Frame: From baseline through Week 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Infliximab | PF-06687234 20 mg + Infliximab
Number analyzed (Participants) | 10 | 10
Participants
  Sitting systolic blood pressure (SBP) < 90 mmHg | 0 | 0
  Increase in Sitting SBP >=30 mmHg | 2 | 0
  Decrease in Sitting SBP >=30 mmHg | 0 | 0
  Sitting diastolic blood pressure (DBP) < 50 mmHg | 0 | 0
  Increase in Sitting DBP >=20 mmHg | 2 | 2
  Decrease in Sitting DBP >=20 mmHg | 3 | 2
  Sitting Pulse Rate < 40 beats/minute | 0 | 0
  Sitting Pulse Rate > 120 beats/minute | 0 | 0

18. Primary Outcome: Number of Participants With Categorical Electrocardiogram (ECG) Data
Description: Twelve (12) lead ECGs were collected. All scheduled ECGs were performed after the participants had rested quietly for at least 10 minutes in a supine position. When the timing of these measurements coincided with a blood collection, the ECG was obtained prior to the nominal time of the blood collection, blood pressure, and pulse rate. ECG data were analyzed as per pre-specified categories. PR=pulse rate; QTc=QT interval corrected for heart rate; QTcF=QTc corrected using Fridericia's formula.
Time Frame: From baseline through Week 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Infliximab | PF-06687234 20 mg + Infliximab
Number analyzed (Participants) | 10 | 10
Participants
  PR Interval >=300 millisecond (msec) | 0 | 0
  Change in PR Interval (%) >=25/50% | 0 | 0
  QRS Complex >=140 msec | 0 | 0
  Change in QRS Complex (%) >=50% | 0 | 0
  QT Interval >=500 msec | 0 | 0
  450 msec ≤ QTcF < 480 msec | 0 | 0
  480 msec <= QTcF < 500 msec | 0 | 0
  QTcF >=500 msec | 0 | 0
  30 msec <= change in QTcF < 60 msec | 0 | 1
  Change in QTcF >=60 msec | 0 | 0

ADVERSE EVENTS:
Time Frame: From the time the participant provided informed consent through Week 22.
Description: All participants who received at least one dose of randomized treatment were included in the analysis for AEs and SAEs.
Arm/Group | Placebo + Infliximab | PF-06687234 20 mg + Infliximab
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/10
Other Adverse Events (participants affected / at risk) | 7/10 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Infliximab (N=10) | PF-06687234 20 mg + Infliximab (N=10)
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Infliximab (N=10) | PF-06687234 20 mg + Infliximab (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Glossitis (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 0 | 2
Fatigue (General disorders) | 0 | 1
Injection site erythema (General disorders) | 0 | 1
Injection site reaction (General disorders) | 0 | 3
Oedema (General disorders) | 0 | 1
Xerosis (General disorders) | 0 | 1
Injection site rash (General disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Onychomycosis (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2
Cardiac murmur (Investigations) | 1 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 2
Stress (Psychiatric disorders) | 0 | 1
Diabetic nephropathy (Renal and urinary disorders) | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 1
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Cushingoid (Endocrine disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated after an interim analysis, due to efficacy being considered unlikely to meet the projected target.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-04-10): https://cdn.clinicaltrials.gov/large-docs/95/NCT03269695/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-02): https://cdn.clinicaltrials.gov/large-docs/95/NCT03269695/SAP_001.pdf